CLINICAL TRIAL: NCT05699135
Title: Treatment Effectiveness of Avelumab First-Line Maintenance Among Canadian Patients With Advanced Urothelial Carcinoma (TRAVELER)
Brief Title: A Study to Learn About the Effect of Avelumab First-Line Maintenance in Canadian People With Advanced Bladder Cancer
Status: Terminated | Type: Observational
Why Stopped: The trial was terminated for strategic reasons. The decision was not based on any safety and/or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B9991053; TRAVELER (Other: Alias Study Number)
Record Dates: First submitted 2022-12-15; First posted 2023-01-26 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Urinary Bladder Neoplasms; Bladder Cancer; Bladder Tumors; Urothelial Carcinoma
Keywords: Bladder Cancer; Bladder Neoplasms; Bladder Tumors; Cancer of Bladder; Cancer of the Bladder; Malignant Tumor of Urinary Bladder; Neoplasms, Bladder; Urinary Bladder Cancer; Metastatic bladder cancer; Locally advanced bladder cancer; Urothelial carcinoma; Locally advanced urothelial carcinoma; Metastatic urothelial carcinoma; avelumab; avelumab maintenance; Canada bladder cancer; Non-interventional study
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Canadian Patients with Advanced Urothelial Carcinoma: Patients with LA/mUC who following 4-6 cycles of platinum chemotherapy and have not progressed, received avelumab, recommended dose of 10mg/kg body weight intravenously administered over 60 minutes every 2 weeks
  Interventions: Drug: Avelumab first-line maintenance

INTERVENTIONS:
Drug: Avelumab first-line maintenance — Patients with LA/mUC who following 4-6 cycles platinum chemotherapy and have not progressed, received avelumab, recommended dose of 10mg/kg body weight, intravenously administered over 60 minutes every 2 weeks

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (called avelumab) for the treatment of advanced bladder cancer.

This study is including participants who:

* Participated in the Canadian avelumab patient support program
* Have been diagnosed with advanced bladder cancer
* Have been treated with platinum-based chemotherapy without their disease progressing All participants in this study have previously received avelumab first-line maintenance for the treatment of their advanced bladder cancer.

Pfizer will examine the experiences of people receiving the study medicine. This will help determine the efficacy and safety of the study medicine for the treatment of bladder cancer.

DETAILED DESCRIPTION:
Avelumab was approved by Health Canada in December 2020 for the maintenance treatment of patients with locally advanced/metastatic urothelial carcinoma (LA/mUC) whose disease has not progressed following first-line (1L) platinum-based chemotherapy. As the urothelial carcinoma treatment landscape evolves with novel indications for previously existing medicines and novel agents entering the market, additional insights are needed to assist in guiding treatment decision making. No observational studies of treatment patterns and outcomes for patients in Canada treated with avelumab first-line maintenance (1LM) have been conducted. The purpose of the current study is to conduct an analysis of patient and disease characteristics and treatment patterns to further elucidate the clinical effectiveness and impact of avelumab 1LM therapy for patients with LA/mUC in Canada.

The primary research objective is to assess effectiveness outcomes in a clinical setting for Canadian patients with LA/mUC treated with avelumab 1LM therapy, specifically overall survival (OS) from the date of avelumab 1LM initiation to the date of death from any cause and progression-free survival (PFS) from the date of avelumab 1LM initiation to the date of progression or death from any cause. Selected secondary objectives include describing treatment patterns, describe AEs explicitly attributed to avelumab among patients with LA/mUC treated with avelumab 1LM and response rates from date of avelumab 1LM initiation, and separately, from the date of chemotherapy initiation, and duration of response (DOR) from date of best overall response in each line of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Canadian avelumab1LM Patient support program (PSP)
* Histologically confirmed diagnosis of stage IV LA/mUC
* No evidence of disease progression following first-line platinum-based chemotherapy
* Receipt of avelumab1LM following 1L platinum-based chemotherapy
* Received the last dose of chemotherapy no more than 10 weeks before entering the PSP
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* ≥6 months of follow-up from initiation of AVE 1LM therapy until study end date, unless the patient has died, with known date of death.

Exclusion Criteria:

* Diagnosed with LA/mUC and enrolled in the PSP, but did not receive avelumab
* Pregnancy at index date
* Participation in an interventional clinical trial at any point during the study period

The index date will be considered as the initiation of index therapy. The index therapy will be considered as the avelumab 1LM treatment after 1L platinum-based chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadian patients histologically diagnosed with stage IV LA/mUC and having participated in the avelumab patient-support program (PSP).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 12 months
  OS from the date of avelumab initiation to the date of death from any cause
Progression-free survival | 12 months
  Progression-free survival from the date of avelumab first-line maintenance initiation to the date of progression or death from any cause

SECONDARY OUTCOMES:
Adverse events explicitly attributed to avelumab | 12 months
  Description of AEs explicitly attributed to avelumab among patients with LA/mUC treated with AVE 1LM
Response rate | 12 months
  Response rate from date of AVE 1LM initiation, and separately, from the date of chemotherapy initiation, and DOR from date of best overall response in each line of therapy
Description of patient characteristics | 12 months
Overall survival from the date of chemotherapy initiation to the date of death from any cause | 12 months
  OS from the date of chemotherapy initiation (prior to AVE 1LM) to the date of death from any cause
Progression-free survival from the date of chemotherapy initiation to the date of progression or death from any cause | 12 months
  PFS from the date of chemotherapy initiation (prior to AVE 1LM) to the date of progression or death from any cause
First-Line therapy description | 12 months
  First-line therapy type, dose, number of cycles, switching and discontinuations
Time to post-diagnostic imaging | 12 months
  Time to post-diagnostic imaging
Time to treatment discontinuation | 12 months
  Time to treatment discontinuation
Time to initiation of AVE 1LM following last dose of chemotherapy | 12 months
  Time to initiation of AVE 1LM following last dose of chemotherapy
Treatment duration of AVE 1LM | 12 months
  Treatment duration of AVE 1LM
Time to next treatment | 12 months
  Time to next treatment
Reasons for treatment discontinuation | 12 months
  Reasons for treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Bayshore Specialty Rx, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991053